CLINICAL TRIAL: NCT01081860
Title: Correlation of Joint Stiffness and Stiffness of the Skin and the Prevelation of Carpal Tunnel Syndrome (CTS)
Brief Title: Stiffness of the Skin and Joints in Relation to Carpal Tunnel Syndrome
Acronym: STIF-CTS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St. Antonius Hospital (Other)
Responsible Party: dr. A.B. Mink van der Molen, department of plastic surgery St Antonius Hospital
Other Study IDs: STIF CTS
Record Dates: First submitted 2010-03-02; First posted 2010-03-05 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; CTS; Skinstiffness; Jointstiffness
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Carpal tunnel syndrome: Patients with carpal tunnel syndrome
- Trigger finger: Patients with trigger fingers
- Dupuytren Contracture: Patients with Dupuytren
- Trauma to the hand: Patients with an acute trauma to the hand

SUMMARY:
The exact etiology of CTS remains yet unknown. A rise in carpal tunnel pressure is well documented, but why this phenomenon occurs is yet unknown in most patients. There is an absolute or relative narrowing of the carpal tunnel, which results in a compression of the median nerve.

The investigators postulate, that a stiffer flexor retinaculum (roof of carpal tunnel) will be less compliant. As a consequence of this stiffer retinaculum the pressure in the carpal tunnel will rise more quickly in stiff patients resulting in CTS-complaints.

A relation between connective tissue composition and joint stiffness is proven. This relationship possibly extends to a relation between stiffness of the skin, joint stiffness and the prevalence of CTS.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Carpal tunnel release OR Trigger finger OR Dupuytren OR an acute trauma to the hand

Exclusion Criteria:

* Hypo-/hyperthyroidism
* Diabetes
* Arthritis
* Pregnancy
* Obesity (BMI >30)
* Anatomical anomalies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients presenting with complaints of:
  * Carpal tunnel syndrome
  * Trigger finger
  * Dupuytren contracture
  * an acute trauma to the hand
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Joint stiffness | In the 1st month
  The active range of motion (elbow, wrist, knee and ankle) is measured with a standard goniometer.
Stiffness of the skin | in the 1st month
  Skinstiffness is measured with a suction cup

SECONDARY OUTCOMES:
Physical activities | In the 1st month
  Boston Questionairre

CONTACTS AND LOCATIONS:
Overall Officials: A.B. Mink van der Molen, dr., Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands